CLINICAL TRIAL: NCT03118843
Title: An Open-Label Study to Evaluate the Safety And Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir Fixed-Dose Combination for 12 Weeks in Subjects Who Participated in a Prior Gilead-Sponsored HCV Treatment Study
Brief Title: Safety And Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir Fixed-Dose Combination for 12 Weeks in Adults Who Participated in a Prior Gilead-Sponsored HCV Treatment Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-4181; 2017-000179-98 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL/VOX (Experimental): SOF/VEL/VOX for 12 weeks
  Interventions: Drug: SOF/VEL/VOX

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg FDC tablet administered orally once daily with food
  Other Names: GS-7997/GS-5816/GS-9857; Vosevi®

SUMMARY:
The primary objectives of this study are to determine the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) fixed-dose combination (FDC) for 12 weeks in participants with chronic hepatitis C virus (HCV) infection with or without cirrhosis, who did not achieve sustained viral response (SVR) after receiving prior treatment in a Gilead-sponsored HCV treatment study of direct-acting antiviral (DAA)-containing regimens.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronically HCV-infected males and non-pregnant/non-lactating females aged 18 years or older who did not achieve sustained virologic response (SVR) in a prior Gilead-sponsored HCV treatment study

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (27):
- United States (17):
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Inland Empire Liver Foundation, Rialto, California
  - Kaiser Permanente, San Diego, California
  - University of Colorado Denver (Leprino Building), Aurora, Colorado
  - Orlando Immunology Center, Orlando, Florida
  - Emory Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Saint Louis University, Gastroenterology & Hepatology, Clinical Research Unit, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center/ New York Presbyterian, New York, New York
  - Center for Liver Diseases, Oakland, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - University of Washington/Harborview Medical Center, Seattle, Washington
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Translational Research Centre, Darlinghurst, New South Wales
- Canada (2):
  - Kay Edmonton Clinic, Edmonton
  - Toronto Centre for Liver Disease (TCLD), Toronto General Hospital, Toronto
- Centre Hospitalier Universitaire de Rouen, Rouen, France
- Germany (2):
  - Leber- and Studienzentrum am Checkpoint, Berlin
  - Universitatsklinikum Bonn, Bonn
- New Zealand (2):
  - Auckland Clinical Studies Ltd, Grafton, Auckland
  - Christchurch Clinical Studies Trust, Ltd, Christchurch
- Kings College Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Result] Ruane P, Strasser SJ, Gane EJ, Hyland RH, Shao J, Dvory-Sobol H, et al. Retreatment with Sofosbuvir/Velpatasvir/Voxilaprevir for 12 weeks is safe and effective for patients who have previously received Sofosbuvir/Velpatasvir or Sofosbuvir/Velpatasvir/Voxilaprevir [Abstract LBO-06]. 16th International Symposium on Viral Hepatitis and Liver Diseases (ISVHLD); 2018 14-17 June; Toronto, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, New Zealand, and Australia. The first participant was screened on 25 April 2017. The last study visit occurred on 19 March 2018.
Pre-assignment Details: 38 participants were screened.
Groups:
- SOF/VEL/VOX: Sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) (400/100/100 mg) fixed-dose combination (FDC) tablet once daily for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL/VOX
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL/VOX: SOF/VEL/VOX (400/100/100 mg) FDC tablet once daily for 12 weeks
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 25
  Race: Black or African American | 5
  Race: Not Disclosed | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 3
  Canada | 2
  United States | 20
  United Kingdom | 1
  Australia | 2
  France | 1
  Germany | 2
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 19
  Genotype 2 | 2
  Genotype 3 | 8
  Genotype 4 | 1
  Genotype 5 | 1
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 3
    CT | 21
    TT | 7
Cirrhosis Status [Count of Participants; unit: Participants]
  Yes | 15
  No | 16
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.56)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 6
  ≥ 800,000 IU/mL | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
percentage of participants | 100.0 [88.8 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to Week 12
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
percentage of participants | 100.0 [88.8 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment
Time Frame: Weeks 2, 4, 8, and 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
percentage of participants
  Week 2 | 51.6 [33.1 to 69.8]
  Week 4 | 96.8 [83.3 to 99.9]
  Week 8 | 100.0 [88.8 to 100.0]
  Week 12 | 100.0 [88.8 to 100.0]

5. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after 2 consecutive HCV RNA < LLOQ), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse: Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Up to Posttreatment Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
percentage of participants | 0

6. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 31
log10 IU/mL
  Change at Week 2: number analyzed (Participants) | 29
  Change at Week 2 | -5.16 (0.560)
  Change at Week 4: number analyzed (Participants) | 30
  Change at Week 4 | -5.34 (0.571)
  Change at Week 8 | -5.34 (0.563)
  Change at Week 12 | -5.34 (0.563)

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to 12 weeks plus 30 days; All-Cause Mortality: Up to Posttreatment Week 12
Description: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL/VOX: SOF/VEL/VOX (400/100/100 mg) fixed-dose combination (FDC) tablet once daily for 12 weeks
Arm/Group | SOF/VEL/VOX
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX (N=31)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX (N=31)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 5
Pain (General disorders) | 2
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Headache (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03118843/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03118843/SAP_001.pdf